CLINICAL TRIAL: NCT06424886
Title: The Effect of Verbal Combined Focus of Attention and Video Instruction Training on Landing Technique and Proprioception in Semi-Professional Female Athletes
Brief Title: The Effect of Different Instruction Trainings in Semi-Professional Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BT-FocusT
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Injury;Sports
Keywords: motor learning; knee valgus; landing biomechanics; proprioception
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: a randomized, controlled, single-blind, prospective study
Who Masked: Outcomes Assessor
Masking Description: Randomization will be done by sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video Instructed Training Group (Experimental): Before the study is conducted, the expert video that will be used for the VI group instructions will be created. The expert video will be created with an athlete with a LESS score of less than 4 and an FPPA of less than 100 who performs a DVJ task in accordance with the instructions. A video recording will be taken of the person designated as an expert performing the DVJ task. The video recording will be used only for the VI group instructions.
  Interventions: Other: Landing error scoring system (LESS)
- Verbal Combined Focus Instructed Training Group (Experimental): It was emphasized that the participants should jump from the 30 cm high box and immediately after landing, jump as high and forward as possible and maintain the final landing stance for 5 seconds. Participants were asked to perform 5 drop vertical jumps and the jumps performed were evaluated. After pretest evaluations were recorded, verbal training group participants performed two training blocks, receiving instructions specific to their group. Participants were given a combined verbal instruction such as "Focus on how hard you push yourself off the ground after the jump and how quickly you straighten your knees during this push", in which internal and external focus directions were given simultaneously. After receiving the instructions, the participants performed 2 drop vertical jumps, 10 times each.
  Interventions: Other: Landing error scoring system (LESS)
- Control Group (Experimental): Participants will be explained how to do the DVJ task in the same way as other groups. Then, after the participants' measurements will be taken, they will start the training blocks without any instructions. Participants will not receive any feedback during training blocks.
  Interventions: Other: Landing error scoring system (LESS)

INTERVENTIONS:
Other: Landing error scoring system (LESS) — Each group will perform two training blocks of 10 drop vertical jumping (DVJ) tasks. Knee joint position sense (KJPS), frontal plane projection angle (FPPA), and Landing Error Scoring System (LESS) assessments will be performed before and after the training blocks, and follow-up assessments will be performed 1 week later. The dominant limb of the participants (the side limb they use when kicking the ball) will be taken into account during the measurement.
  Other Names: drop vertical jump landing task; frontal plane projection angle (FPPA); knee joint position sense (KJPS)

SUMMARY:
Feedback is implanted into workouts to prevent lower extremity injuries. There are different studies where external focus and internal focus feedback were found to be superior. The main purpose of this study is to investigate the effects of training on vertical jump landing technique by comparing a verbal training group that receives instructions with an external focus of attention and an internal focus of attention combined, a visual training group with video instructions, and a control group in female athletes with knee valgus. It is also to examine whether possible beneficial results are still present in the retention test performed one week after the test session. The secondary aim of our study is to examine the effect of the training provided on knee joint position sense.

DETAILED DESCRIPTION:
Approximately 70% of lower extremity injuries occur during non-contact, single-leg landings, and jumping to the ground is a common injury mechanism in both genders. Additionally, female athletes have higher injury rates compared to men, potentially due to anatomical differences of the lower kinematic chain. Events in which athletes experience non-contact ACL injuries generally show many common biomechanical features such as increased ground reaction forces during single-leg landing, decreased joint flexion in the sagittal plane of the ankle, knee, hip and trunk, as well as increased knee internal rotation angles. Another critical ACL injury risk factor is performing a secondary task during sharp deceleration movements. Current rehabilitation programs focus on neuromuscular training programs to prevent adverse movement patterns and increase proper movement control. However, there is still a need to increase the effectiveness of these neuromuscular training programs to have a more significant impact on ACL injury rates. Therefore, the use of motor learning strategies and neuromuscular training programs with adequate and correct techniques in the rehabilitation of athletes should still be investigated.

There are various approaches to motor learning. One of the best-known approaches is the cognitive approach, where the athlete reaches the automation stage by receiving feedback and repeating the model technique as often as possible. The common denominator of motor learning strategies is the use of explicit instructions and feedback regarding desired landing positions. Instructions for the implementation of movements in rehabilitation programs aim to improve performance and motor learning. These instructions may address the action outcome or the course of action. There are many studies showing that feedback training changes jump landing biomechanics. In line with the results of these studies, using feedback techniques, especially to reduce the vertical ground reaction force and increase the knee flexion angle during landing from a jump, can reduce the stress and risk of injury in the lower extremity.

Motor skills can be learned with an internal focus of attention or with an external focus of attention. Although the difference in these instructions may seem insignificant, externally focused education; has been shown to result in better performance, retention, transfer, and greater movement automaticity. The main purpose of this study is to investigate the effects of training on vertical jump landing technique by comparing a verbal training group that receives instructions with an external focus of attention and an internal focus of attention combined, a visual training group with video instructions, and a control group in female athletes with knee valgus. It is also to examine whether possible beneficial results are still present in the retention test performed one week after the test session. The secondary aim of our study is to examine the effect of the training provided on knee joint position sense.

ELIGIBILITY:
Inclusion Criteria:

* Being female
* Being between the ages of 18-24
* Body mass index being between 18.5 kg/m2 and 25 kg/m2
* Becoming a minor league basketball or volleyball player
* Volunteers must not have suffered any trunk or lower extremity injuries in the last 6 months before participation in the study.
* Having a frontal plane projection angle greater than 100 during the single-leg squat test

Exclusion Criteria:

* • Having experienced a trunk or lower extremity injury in the last 6 months before the date of study

  * Having a history of fracture or dislocation in the lower extremity
  * Having suffered from back pain in the past years
  * Having a musculoskeletal system abnormality
  * Being unable to perform functional tasks (visual, auditory, vestibular or neurological impairment)
  * Being pregnant
  * Having malignancy and metabolic diseases

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Landing Error Scoring System (LESS) Measurement | baseline, immediately after the intervention, one week after the baseline
  Two standard video cameras capture the frontal plane and sagittal plane view of each subject as they perform the test procedures (jumping from 30 cm height box). The participant's LESS score represents excellent (LESS score <4), good (LESS score >4 to 5), fair (LESS score >5 to 6) and poor (LESS score >6) jumping technique.

SECONDARY OUTCOMES:
Frontal Plan Projection Angle (FPPA) Measurement | baseline, immediately after the intervention, one week after the baseline
  During the frontal plane projection angle (FPPA) measurement, a straight line will be drawn from the anterior superior spina iliaca along the femur to the midpoint of the patella, and the midpoint of the ankle will be determined as the reference point by a straight line drawn from the midpoint of the patella. Participants will stand with their feet aligned in the sagittal plane and their arms crossed across their chests. By prior instruction, subjects will be asked to squat up to 60º knee flexion in a controlled manner without losing their balance, before returning to the starting position. Digital recordings of the frontal plane will be made while individuals perform a single-leg squat test at 60º knee flexion 3 times. The FPPA degree is measured from the medial aspect of the knee and calculated by subtracting 360. FPPA of 195° and above will be considered pathological.
Knee Joint Position Sense (KJPS) Measurement | baseline, immediately after the intervention, one week after the baseline
  Participants are initially placed in a sitting position in 90° knee flexion. Participants' eyes are covered with a mask to block visual input. The smartphone that will perform the measurement is fixed to the participants' lower limb (15 cm from the apex of the fibular head) with a Velcro strap. From the starting position (90 knee flexion), the participants' knee is placed by the researcher at a target joint angle of 45. Participants actively hold the knee at the 45 target joint angle for five seconds to understand the exact angle of the knee. After these five seconds, the participants actively return their knee to the starting position and the researcher shows the target angle to the participant three times. With the command given by the researcher, the participants are directed to extend their knees as close as possible to the target joint angle without any external stimulation or assistance. Participants perform 3 trials and try to maintain the estimated position for 3 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, PT, PhD, Study Director — Bahcesehir University, Faculty of Health Sciences, Department of Physiotherapy; Büşra Tamgüç, PT, Principal Investigator — Bahcesehir University, Graduate Education Institute
Locations (1):
- Istanbul Panterler Sports Club, Kağıthane, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Tamguc B, Pisirici P. The Effect of Verbal Combined Focus of Attention and Video Instruction Training on Knee Valgus and Landing Technique in Semiprofessional Female Athletes. Orthop J Sports Med. 2025 Apr 4;13(4):23259671251326454. doi: 10.1177/23259671251326454. eCollection 2025 Apr. PMID 40291630